CLINICAL TRIAL: NCT03626831
Title: Randomized, Double-blind, Placebo Controlled, Parallel-group, Prospective Clinical Study to Analyse the Effect of Evolocumab on Vascular Function
Brief Title: Effect of Evolocumab on Vascular Function
Acronym: EVO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Principal Investigator, Roland E. Schmieder, Full Professor of Medicine, University of Erlangen-Nürnberg Medical School
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CRC2017EVO
Record Dates: First submitted 2018-08-08; First posted 2018-08-13 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2023-07

CONDITIONS: Atherosclerotic Cardiovascular Disease
Keywords: CVD; LDL; heart failure; PCSK9
MeSH Terms: conditions — Atherosclerosis; Heart Failure

STUDY DESIGN:
Intervention Model Description: randomized (1:1), prospective, double-blind, placebo controlled, parallel-group
Who Masked: Participant, Care Provider, Investigator
Masking Description: double blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment (Active Comparator): Baseline vascular function parameters will be obtained and the patient will be given an SC injection of the study drug by Evolocumab Prefilled Syringe (1x SC 420 mg evolocumab).
  Interventions: Drug: Evolocumab Prefilled Syringe
- Placebo (Placebo Comparator): Baseline vascular function parameters will be obtained and the patient will be given an SC injection of Placebos (1x SC Placebo).
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Evolocumab Prefilled Syringe — Injection of study drug
  Arms: Treatment
Drug: Placebos — Injection of placebo
  Arms: Placebo

SUMMARY:
This is a phase IV, randomized (1:1), prospective, double-blind, placebo controlled, parallel-group, single center study at the Clinical Research Unit (CRC) of the Department of Nephrology and Hypertension, with its two separate locations:

* Nürnberg, Kreuzburger Str. 2, 90471 Nürnberg, and
* Erlangen, Ulmenweg 18, 91054 Erlangen

The results of this study provide strong support for the concept that it is lower LDL-C levels that is key to achieving better outcomes, and that it is possible to achieve these on top of statin therapy (despite the much debated potential "pleiotropic" effects of statins).

At least 65 patients will be randomized (1:1) and included (informed consent) in order to obtain 58 fully evaluable subjects (29 with evolocumab, 29 with placebo).

Patients will be simultaneously recruited from investigator's outpatient clinics, referring physicians, and advertisement in local newspapers, and social media. Those patients that appear to potentially fulfill the inclusion criteria will be invited to a screening visit. After providing informed consent, patients will be tested for inclusion/exclusion criteria and for feasibility of vascular measurements (in particular to ensure that adequate imaging of the brachial artery is possible). Patients will provide a blood sample for laboratory testing. If the patient then fulfills inclusion criteria and in the absence of exclusion criteria, the patient will be enrolled into the trial, and the study visits will be scheduled. Randomization will take place at the latest one day prior to the study visit 2 (e.g. at the latest at visit 2a).

At visit 2, baseline vascular function parameters will be obtained and the patient will be given an SC injection of the study drug (either SC 420 mg evolocumab or SC placebo). At visit 4, the second injection of study drug will be administered. After 1, 4 and 8 weeks of treatment (visits 3, 4 and 5), testing of vascular function will be repeated. At visit 6, a final close out visits will be performed to gather additional safety information.

DETAILED DESCRIPTION:
The recently published IMPROVE-IT trial was the first to demonstrate that in high-risk patients, reduction of low density cholesterol (LDL-C) beyond current treatment goals by addition of ezetimibe to statin therapy leads to a further improvement of cardiovascular (CV) outcomes. The results of this study provide strong support for the concept that it is lower LDL-C levels that is key to achieving better outcomes, and that it is possible to achieve these on top of statin therapy (despite the much debated potential "pleiotropic" effects of statins). However, ezetimibe has only limited ability to reduce LCL-C further (-24% lower compared with statin alone in the IMPROVE-IT trial). Proprotein convertase subtilisin/kexin type 9 (PCSK9) inhibition is a new treatment paradigm for hypercholesterolemia. The normal function of PCSK9 is to bind to the low density cholesterol (LDL-C) receptor, and to promote its lysosomal destruction in the hepatocyte. Thus, inhibition of PCSK9 protects the LDL-C receptor from lysosomal destruction, resulting in increased recirculation of the LDL-C receptor to the hepatocyte cell surface, and as a consequence, increased hepatic uptake and lower circulating levels of LDL-C.

The PCSK9 inhibitor evolocumab has been approved in 2015 for the treatment of patients with homocygote familial hypercholesterolemia (FH), as well as for treatment of patients with heterocygote familial or non-familial hypercholesterolemia in which target LDL-C levels cannot be achieved by standard cholesterol-lowering therapy, or who are statin-intolerant. Evolocumab achieves a reduction in LDL-C regardless of background therapy in the order of 50-70% (including those on a statin). This therapy substantially increases the number of patients achieving lower LCL-C target levels. Recently, the results of a large prospective study (FOURIER) in 27.500 patients at high CV risk have been published. This study showed that evolocumab lowered LDL cholesterol in patients already on optimized lipid lowering therapy including a statin to a median of 30 mg per deciliter and substantially reduced CV events (hazard ratio 0.85, confidence interval 0.79 to 0.92; P<0.001). However, the mechanisms mediating the improvement of CV outcomes under therapy with evolocumab are unclear at present.

Intact function of the endothelium is a key component of vascular health. Conversely, impaired endothelial function has been linked with increased future CV event rates. Intact endothelium has many protective and anti-atherosclerotic effects on the vasculature. At least in part, these protective effects are due to endothelial release of nitric oxide (NO). A well-established and non-invasive method of assessing endothelial function in humans is by measurement of flow-mediated vasodilation (FMD). In addition, recent evidence suggests concurrent assessment of low flow-mediated vasoconstriction (L-FMC) improves characterization of underlying CV and coronary disease compared with each parameter alone. Further, endothelial function has been found to impact large artery function. Endothelial dysfunction leads to vasoconstriction, greater peripheral wave reflection and arterial stiffness, and as a consequence, augmentation of central (aortic) systolic blood pressure (BP). This is of prognostic relevance, since aortic stiffness (e.g. determined by pulse wave velocity [PWV]), central systolic BP (cSBP) and central BP augmentation have been identified as strong and independent predictors of CV events in several patient cohorts. Exciting technical developments of recent years have now made the ambulatory (24-h) measurement of arterial stiffness possible.

The investigator group has been amongst the first to show that statin treatment improves endothelial function in patients with elevated LDL-C, which at least in part serves to explain the beneficial effects of statins on CV outcomes. The investigator Group was also able to show that an improvement in endothelial function during statin therapy is linked with an improvement of pulse wave reflection. Rapid improvement of endothelial and large artery function is considered to be particularly important in patients at high CV risk, such as those that have suffered a recent CV event. The investigator Group hypothesize that the beneficial effects of evolocumab, such as recently demonstrated in the FOURIER trial, are linked to a rapid improvement of endothelial and large artery function, even in patients already on optimized lipid lowering therapy including a statin. Of note, improvement of basal NO activity in the renal circulation and NO-dependent vasodilation of the peripheral vasculature occurs already 3 days after initiating treatment of statins. In the current study we focus on FMD of the brachial artery as the primary objective parameter. This parameter, which is widely accepted as an integrated measure of vascular function, is partly dependent on endothelial NO production. These data would help to explain the results of IMPROVE-IT and FOURIER, and add to the evidence that it is lower cholesterol levels that matter most for CV outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent in written form
* Male or female 40 - 80 years
* History of clinically evident atherosclerotic cardiovascular disease as evidenced by ANY of the following:
* diagnosis of coronary artery disease as evidenced by acute coronary syndrome, myocardial infarction (MI), coronary stent implantation, coronary stenosis ≥50% by coronary angiography
* diagnosis of non-hemorrhagic stroke or transient ischemic attack (TIA)
* symptomatic peripheral arterial disease (PAD), as evidenced by intermittent claudication with ankle-brachial index (ABI) < 0.85, or peripheral arterial revascularization procedure, or amputation due to atherosclerotic disease, or artery stenosis ≥50% by angiography
* Fasting LDL-C ≥ 70 mg/dL (≥ 1.8 mmol/L) or non-HDL-C ≥ 100 mg/dL (≥ 2.6mmol/L) on optimized background lipid lowering therapy (please see Appendix 14.3.)
* Stable background lipid lowering therapy for at least 4 weeks (please see Appendix 14.3)
* Most recent fasting triglycerides ≤ 400 mg/dL (4.5 mmol/L) by central laboratory before randomization

Exclusion Criteria:

* Inability to image the brachial artery and to perform FMD
* Subjects with statin intolerance
* Known or suspected homozygous familial hypercholesterolemia (FH)
* Subject must not be randomized within 4 weeks of their most recent MI or stroke
* NYHA class III or IV, or last known left ventricular ejection fraction < 30%
* Atrial fibrillation
* Known hemorrhagic stroke at any time
* Uncontrolled or recurrent ventricular tachycardia
* Planned or expected cardiac surgery or revascularization within 3 months after randomization
* Uncontrolled hypertension defined as sitting pSBP > 180 mmHg or pDBP > 110 mmHg
* Use of cholesteryl ester transfer protein (CETP) inhibition treatment, mipomersen, or lomitapide within 12 months prior to randomization. Fenofibrate therapy must be stable for at least 6 weeks prior to final screening at a dose that is appropriate for the duration of the study in the judgment of the investigator. Other fibrate therapy (and derivatives) are prohibited
* Prior use of PCSK9 inhibition treatment other than evolocumab or use of evolocumab < 12 weeks prior to final lipid screening
* Untreated or inadequately treated hyperthyroidism or hypothyroidism as defined by thyroid stimulating hormone (TSH) < lower limit of normal (LLN) or > 1.5 times the upper limit of normal (ULN), respectively, and free thyroxine (T4) levels that are outside normal range at final screening
* Severe renal dysfunction, defined as an estimated glomerular filtration rate (eGFR) < 30 mL/min/1.73m2 at final screening
* Active liver disease or hepatic dysfunction, defined as serum Glutamate-Oxaloacetate-Transaminase (SGOT) or serum Glutamate-Pyruvate-Transaminase (SGPT)> 3 times the ULN as determined by central laboratory analysis at final screening
* Recipient of any major organ transplant (eg, lung, liver, heart, bone marrow, renal)
* Personal or family history of hereditary muscular disorders
* LDL or plasma apheresis within 12 months prior to randomization
* Severe, concomitant non-CV disease that is expected to reduce life expectancy to less than 3 years
* Creatinine Kinase (CK) > 5 times the ULN at final screening
* Known major active infection or major hematologic, renal, metabolic, gastrointestinal or endocrine dysfunction in the judgment of the investigator
* Malignancy (except non-melanoma skin cancers, cervical in-situ carcinoma, breast ductal carcinoma in situ, or stage 1 prostate carcinoma) within the last 10 years
* Subject has received drugs via a systemic route that have known major interactions with background statin therapy (see Appendix 14.4.) within 1 month prior to randomization or is likely to require such treatment during the study period
* Currently enrolled in another investigational device or drug study, or less than 30 days since ending another investigational device or drug study(s), or less than 5 fold of half-live time of the investigational drug, or receiving other investigational agent(s)
* Female subject who has either (1) not used acceptable method(s) of birth control for at least 1 month prior to screening or (2) is not willing to use such a method during treatment with IP and for an additional 15 weeks after the end of treatment with IP, unless the subject is sterilized or postmenopausal;

  * menopause is defined as 12 months of spontaneous and continuous amenorrhea in a female ≥ 55 years old or 12 months of spontaneous and continuous amenorrhea with a follicle-stimulating hormone (FSH) level > 40 IU/L (or according to the definition of "postmenopausal range" for the laboratory involved) in a female < 55 years old unless the subject has undergone bilateral oophorectomy
  * acceptable methods of preventing pregnancy include not having intercourse, birth control pills, injections, implants, or patches, intrauterine devices (IUDs), tubal ligation/occlusion, sexual activity with a male partner who has had a vasectomy, condom or occlusive cap (diaphragm or cervical/vault caps) used with spermicide
* Subject is pregnant or breast feeding, or planning to become pregnant or to breastfeed during treatment with IP and/ or within 15 weeks after the end of treatment with IP
* Known sensitivity to any of the active substances or their excipients to be administered during dosing
* Subject likely to not be available to complete all protocol-required study visits or procedures, to the best of the subject's and investigator's knowledge

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2019-04-04 (Actual); Primary Completion 2021-04-15 (Actual); Study Completion 2021-07-12 (Actual)

PRIMARY OUTCOMES:
Percent change of FMD | 8 weeks
  Percent change of FMD (UNEX EF) after 8 weeks of treatment from baseline

SECONDARY OUTCOMES:
Absolute change of FMD (UNEX EF) | 8 weeks
  Absolute change of FMD (UNEX EF) after 8 weeks of treatment from baseline
Absolute change of L-FMC | 8 weeks
  Absolute change of L-FMC after treatment from baseline and across all visits
Percent change of L-FMC | 8 weeks
  Percent change of L-FMC after treatment from baseline and across all visits
Absolute change of combined FMD+L-FMC (UNEX EF) | 8 weeks
  Absolute change of combined FMD+L-FMC (UNEX EF) after treatment from baseline and across all visits.
Percent change of combined FMD+L-FMC (UNEX EF) | 8 weeks
  Percent change of combined FMD+L-FMC (UNEX EF) after treatment from baseline and across all visits.

CONTACTS AND LOCATIONS:
Overall Officials: Roland E Schmieder, MD, Principal Investigator — University Hospital Erlangen
Locations (1):
- Clinical Research Center, Department of Nephrology and Hypertension, University of Erlangen-Nuremberg, Erlangen, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gunes-Altan M, Bosch A, Striepe K, Schiffer M, Achenbach S, Schmieder RE, Kannenkeril D. Endothelial function in high-risk patients with ezetimibe therapy. J Clin Lipidol. 2025 Sep-Oct;19(5):1364-1373. doi: 10.1016/j.jacl.2025.07.001. Epub 2025 Jul 9. PMID 40813220